CLINICAL TRIAL: NCT00402688
Title: A Multicenter, Double-Blind, Phase 3B Study to Compare the Safety and Clinical Efficacy of Levofloxacin in 750mg for 2 Weeks and Levofloxacin 750mg for 3 Weeks to That of Levofloxacin 500mg for 4 Weeks in the Treatment of Chronic Prostatitis
Brief Title: An Effectiveness and Safety Study for Levofloxacin in Chronic Prostatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR012103; CR012103 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Prostatitis
Keywords: Chronic Prostatitis; Prostatitis; levofloxacin; Levaquin
MeSH Terms: conditions — Prostatitis | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 001 (Active Comparator): levofloxacin 750mg tablet once daily for 2 weeks followed by 2 weeks of placebo.
  Interventions: Drug: levofloxacin
- 002 (Active Comparator): levofloxacin 750mg tablet once daily for 3 weeks followed by 1 week of placebo.
  Interventions: Drug: levofloxacin
- 003 (Active Comparator): levofloxacin 500mg tablet once daily for 4 weeks.
  Interventions: Drug: levofloxacin

INTERVENTIONS:
Drug: levofloxacin — 750mg tablet once daily for 2 weeks followed by 2 weeks of placebo.
  Arms: 001
Drug: levofloxacin — 750mg tablet once daily for 3 weeks followed by 1 week of placebo.
  Arms: 002
Drug: levofloxacin — 500mg tablet once daily for 4 weeks.
  Arms: 003

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of levofloxacin 750 mg for 2 weeks or 750 mg for 3 weeks, compared to levofloxacin 500 mg for 4 weeks in the treatment of chronic prostatitis.

DETAILED DESCRIPTION:
The optimal duration of treatment for chronic prostatitis remains unclear. Historically, therapy for chronic prostatitis with other classes of antibacterials resulted in poor outcomes and prolonged time taking the medication. Levofloxacin belongs to the quinolone class of antibacterials and has been used to treat chronic prostatitis with 500mg of levofloxacin taken orally once a day for 4 weeks. This multicenter, double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), randomized (patients are assigned different treatments based on chance) study is designed to see if giving levofloxacin at a higher dose for shorter periods of time is safe and effective in treating chronic prostatitis. Safety analyses will involve the examination of the incidence, severity, and type of adverse events and changes in physical findings including vital signs and clinical laboratory tests. Patients will receive one of the following three dosing options: levofloxacin 750 mg orally administered once-a-day for 2 weeks followed by placebo once-a-day for two weeks for a total of 4 weeks, or levofloxacin 750 mg orally once-a-day for 3 weeks followed by placebo once-a-day for one week for a total of 4 weeks, or levofloxacin 500 mg orally once-a-day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males 40 years of age or older
* A clinical diagnosis of chronic prostatitis as evidenced by the following two criteria: 1. Clinical signs and symptoms of prostatitis including a soft, tender prostate without noticeable nodularity with one or more of the following signs or symptoms: painful or difficult urination, suprapubic discomfort, painful ejaculation, low back pain, perineal discomfort, urinary frequency, urinary urgency or hesitancy, decreased urinary stream, urinary retention, pain on digital rectal examination, perineal tenderness or pain, fever, chills. 2. A history of chronic prostatitis as defined as: symptomatic prostatitis - a clinical diagnosis of prostatitis having been made for at least one previous episode that lasted four weeks, or two or more episodes during the previous twelve months.

Exclusion Criteria:

* Any condition which may interfere with the evaluation of study drug including transurethral prostatectomy within six months of enrollment, the presence of a permanent transurethral catheter or a history of cystostomy or nephrostomy
* Taking hormone therapy
* Known prostatic carcinoma
* Allergy to levofloxacin, ofloxacin, ciprofloxacin, or other members of the quinolone class of antibacterials.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (39):
- United States (39):
  - Birmingham, Alabama
  - Homewood, Alabama
  - Anchorage, Alaska
  - Hot Springs, Arkansas
  - Fresno, California
  - San Diego, California
  - Denver, Colorado
  - New Britain, Connecticut
  - New Smyrna Beach, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Plantation, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Columbus, Georgia
  - Roswell, Georgia
  - Jeffersonville, Indiana
  - Des Moines, Iowa
  - Shreveport, Louisiana
  - Greenbelt, Maryland
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Marlton, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - Kingston, New York
  - New York, New York
  - Orchard Park, New York
  - Poughkeepsie, New York
  - Staten Island, New York
  - Salisbury, North Carolina
  - Columbus, Ohio
  - Bethany, Oklahoma
  - Allentown, Pennsylvania
  - Bala-Cynwyd, Pennsylvania
  - State College, Pennsylvania

REFERENCES:
- [Derived] Paglia M, Peterson J, Fisher AC, Qin Z, Nicholson SC, Kahn JB. Safety and efficacy of levofloxacin 750 mg for 2 weeks or 3 weeks compared with levofloxacin 500 mg for 4 weeks in treating chronic bacterial prostatitis. Curr Med Res Opin. 2010 Jun;26(6):1433-41. doi: 10.1185/03007991003795030. PMID 20394471
- See also: An Effectiveness and Safety Study for Levofloxacin in Chronic Prostatitis. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=62&filename=CR012103_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Levofloxacin 750mg for 2 Weeks: levofloxacin, 750mg tablet once daily for 2 weeks followed by 2 weeks of placebo.
- Levofloxacin 750mg for 3 Weeks: levofloxacin, 750mg tablet once daily for 3 weeks followed by 1 week of placebo.
- Levofloxacin 500mg for 4 Weeks: levofloxacin, 500mg tablet once daily for 4 weeks.
Period: Overall Study
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Started | 81 | 81 | 80
Completed | 60 | 65 | 65
Not Completed | 21 | 16 | 15
Not completed — Adverse Event | 12 | 9 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lack of Efficacy | 4 | 4 | 5
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Culture Show Fluoroquinolone Resistance | 0 | 1 | 0
Not completed — Urine Cult. Yield Resistant to Levaquin | 0 | 0 | 1
Not completed — Patient Left Town and Forgot Medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks | Total
Number analyzed (Participants) | 81 | 81 | 80 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 65 | 71 | 65 | 201
  >=65 years | 16 | 10 | 15 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 81 | 81 | 80 | 242

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success
Description: Defined as cured or improved. Response is based on the resolution of signs and symptoms at post-therapy.
Time Frame: Posttherapy Visit (Study Day 33-36)
Population: Modified Intent to Treat (mITT)
Measure: Number; unit: Participants
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Number analyzed (Participants) | 73 | 74 | 75
Participants | 46 | 48 | 52
Statistical Analysis 1: Comparison: Levofloxacin 750mg for 2 Weeks vs Levofloxacin 500mg for 4 Weeks; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is a risk difference of 0.2; Risk Difference (RD) = 0.063, 95% CI [-0.089 to 0.215] — Difference in success rates (levofloxacin 500mg for 4 weeks minus levofloxacin 750mg for 2 weeks )
Statistical Analysis 2: Comparison: Levofloxacin 750mg for 3 Weeks vs Levofloxacin 500mg for 4 Weeks; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is a risk difference of 0.2; Risk Difference (RD) = 0.045, 95% CI [-0.106 to 0.195] — Difference in success rates (levofloxacin 500mg for 4 weeks minus levofloxacin 750mg for 3 weeks)

2. Secondary Outcome: Symptom Relief (Resolved)
Description: Participants With Resolution of Prostatitis Signs and Symptoms; Resolution is defined as symptoms present (mild, moderate or severe) at Screening/Admission and absent (none) at the Posttherapy evaluation.
Time Frame: Posttherapy Visit (Study Day 33-36)
Population: Modified Intent to Treat (mITT)
Measure: Number; unit: Participants
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Number analyzed (Participants) | 73 | 74 | 75
Participants
  Dysuria (n=35, 43, 42) | 23 | 29 | 27
  Suprapubic discomfort (n=41, 36, 45) | 24 | 19 | 30
  Painful ejaculation (n=32, 39, 34) | 17 | 23 | 20
  Low back pain (n=43, 44, 44) | 20 | 22 | 26
  Perineal discomfort (n=40, 42, 50) | 20 | 19 | 29
  Frequency (n=58, 63, 62) | 29 | 24 | 30
  Urgency (n=48, 52, 58) | 20 | 28 | 35
  Hesitancy (n=37, 39, 54) | 19 | 16 | 38
  Decreased urinary stream (n=50, 47, 52) | 24 | 21 | 30
  Urinary retention (n=24, 26, 27) | 13 | 13 | 17
  Pain on digital rectal examination (n=60, 59, 61) | 30 | 30 | 42
  Perineal tenderness or pain (n=44, 38, 43) | 28 | 24 | 28
  Chills (n=4, 5, 7) | 3 | 3 | 7
  Other (n=5, 8, 8) | 1 | 5 | 5
  Fever (n=3, 2, 1) | 2 | 2 | 1

3. Secondary Outcome: Clinical Success (Non-Relapse) or Failure (Relapse)
Description: Number of Clinical Successes or Failures at the 6-Week Poststudy Telephone Contact for Participants Cured/Improved at the Posttherapy Visit
Time Frame: Poststudy Telephone contact at 6 weeks
Population: Modified Intent-to-Treat Population (mITT) (Participants Cured/Improved at the Posttherapy Visit)
Measure: Number; unit: participants
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Number analyzed (Participants) | 46 | 48 | 52
participants
  Clinical Success | 38 | 32 | 44
  Failure | 3 | 12 | 5
  Unable to Evaluate | 0 | 1 | 1
  Missing | 5 | 3 | 2

4. Secondary Outcome: Clinical Success (Non-Relapse) or Failure (Relapse)
Description: Number of Clinical Successes or Failures at 3 Month Poststudy Telephone Contact for Participants Cured/Improved at the Posttherapy Visit
Time Frame: Poststudy Telephone contact at 3 Months
Population: Modified Intent to Treat (mITT) (Participants Cured/Improved at the Posttherapy Visit)
Measure: Number; unit: Participants
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Number analyzed (Participants) | 46 | 48 | 52
Participants
  Clinical Success | 30 | 24 | 38
  Failure | 8 | 6 | 4
  Unable to Evaluate | 0 | 1 | 1
  Missing | 8 | 17 | 9

5. Secondary Outcome: Clinical Success (Non-Relapse) or Failure (Relapse)
Description: Number of Clinical Successes or Failures at the 6-month Poststudy Telephone Contact For Participants Cured/Improved at the Posttherapy Visit
Time Frame: Poststudy Telephone Contact at 6 Months
Population: Modified Intent to Treat (mITT) (Participants Cured/Improved at the Posttherapy Visit)
Measure: Number; unit: Participants
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Number analyzed (Participants) | 46 | 48 | 52
Participants
  Clinical Success | 19 | 19 | 31
  Failure | 10 | 4 | 6
  Unable to Evaluate | 1 | 1 | 1
  Missing | 16 | 24 | 14

6. Secondary Outcome: Total NIH-CPSI Score
Description: National Institute of Health-Chronic Prostatitis Symptom Index numerically rates a total score (0-43) where 0 indicates no symptoms across any of the domains (pain or discomfort, urination, quality of life).
Time Frame: Screening/Admission, On-Therapy, Week 3, Week 4, Posttherapy (Study Day 33-36)
Population: Modified Intent to Treat (mITT)
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Number analyzed (Participants) | 73 | 74 | 75
Score on a scale
  Screening/Admission (n=73, 74, 75) | 11.8 [2 to 27] | 12.0 [3 to 27] | 12.9 [3 to 27]
  On-Therapy (n=70, 70, 73) | 7.2 [0 to 22] | 6.6 [0 to 19] | 6.9 [0 to 19]
  Week 3 (Visit 2) (n=62, 65, 68) | 6.5 [0 to 24] | 6.5 [0 to 21] | 5.6 [0 to 24]
  Week 4 (Visit 3) (n=53, 57, 61) | 5.1 [0 to 19] | 4.9 [0 to 17] | 4.5 [0 to 25]
  Posttherapy (Visit 4) (n=70, 71, 71) | 5.4 [0 to 24] | 5.0 [0 to 21] | 4.6 [0 to 22]

ADVERSE EVENTS:
Arm/Group | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Serious Adverse Events (participants affected / at risk) | 2 | 1 | 0
Other Adverse Events (participants affected / at risk) | 43 | 42 | 38
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Syncope (General disorders) | 1/81 | 0/81 | 0/80
Coronary Artery Disorder (Vascular disorders) | 1/81 | 0/81 | 0/80
Depression (Psychiatric disorders) | 0/81 | 1/81 | 0/80
Hallucination (Psychiatric disorders) | 0/81 | 1/81 | 0/80
Suicidal Ideation (Psychiatric disorders) | 0/81 | 1/81 | 0/80
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Levofloxacin 750mg for 2 Weeks | Levofloxacin 750mg for 3 Weeks | Levofloxacin 500mg for 4 Weeks
Chest Pain (General disorders) | 3/81 | 0/81 | 2/80
Fever (General disorders) | 3/81 | 3/81 | 1/80
Back Pain (General disorders) | 2/81 | 2/81 | 1/80
Pain (General disorders) | 1/81 | 5/81 | 2/80
Fatigue (General disorders) | 0/81 | 1/81 | 2/80
Oedema Peripheral (General disorders) | 0/81 | 1/81 | 2/80
Hypertension (Cardiac disorders) | 0/81 | 2/81 | 1/80
Dizziness (Nervous system disorders) | 9/81 | 3/81 | 2/80
Headache (Nervous system disorders) | 3/81 | 4/81 | 3/80
Nausea (Gastrointestinal disorders) | 8/81 | 6/81 | 2/80
Diarrhoea (Gastrointestinal disorders) | 5/81 | 5/81 | 5/80
Constipation (Gastrointestinal disorders) | 4/81 | 1/81 | 2/80
Abdominal Pain (Gastrointestinal disorders) | 3/81 | 1/81 | 6/80
Dyspepsia (Gastrointestinal disorders) | 3/81 | 1/81 | 1/80
Myalgia (Musculoskeletal and connective tissue disorders) | 4/81 | 2/81 | 2/81
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/81 | 3/81 | 0/80
Skeletal Pain (Musculoskeletal and connective tissue disorders) | 3/81 | 1/81 | 1/80
Fascitis Plantar (Musculoskeletal and connective tissue disorders) | 2/81 | 0/81 | 0/80
Insomnia (Psychiatric disorders) | 5/81 | 2/81 | 3/80
Penis Disorder (Reproductive system and breast disorders) | 0/81 | 2/81 | 0/80
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0/81 | 1/81 | 2/80
Rash (Skin and subcutaneous tissue disorders) | 1/81 | 0/81 | 2/80
Sweating Increased (Skin and subcutaneous tissue disorders) | 0/81 | 2/81 | 2/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less